CLINICAL TRIAL: NCT04326972
Title: Diagnostic Value of Chest Ultrasound in Detecting Causes of Radiological Opacities in Comparison to CT Scan Among Children at Assiut University Children Hospital
Brief Title: Diagnostic Value of Chest Ultrasound in Pediatrics Lung Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dhekra Ashour Aboud Salem, M.S.C, Assiut University
Other Study IDs: chest ultrasound in pediatrics
Record Dates: First submitted 2020-03-27; First posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Lung Diseases
MeSH Terms: conditions — Lung Diseases | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ultrasound — • All patients with inclusion criteria do for them chest ultrasound .

SUMMARY:
To evaluate the accuracy of chest ultrasound for diagnosis of different lung lesions in comparison to the gold standard among children.

DETAILED DESCRIPTION:
Lung disease are the most common condition in pediatrics and also the primary cause of death among children less than 5 years old(Chen Shui-Wen et al.,2015).

Chest X ray consider as the first line to evalute the chest disease (Kim O et al. ,2000), in identified the pulmonary opacities (Ozkaya A et al., 2018),but there is limitation in the interpretation of the location and nature of an area of increase opacity on chest radiographs particularly in young infants with varied configuration of thymus and differentiation between pulmonary , pleural and mediastinal lesions is not always easy(Barillari A et al .,2011),so the thoracic computed tomography is recommended as diagnostic gold standard to follow up pediatric chest X ray opacities and masses(Lameh A et al. ,2019),but not consider as first line of radiological evaluation because each chest computed tomography gives to patient an effective dose of eight msv equivalent to four hundred chest X ray (Prithviraj D.,2014), also high cost ,and longe waiting times for imaging (Lameh A et al .,2019).

Chest sonography consider as first line investigation in evaluation of diaphragmatic ,pleural and chest wall lesions due to lack of superficial adipose tissue in pediatric patients (Goh Y, et al. ,2016),but undervalued for lungs lesion for many years ,because the ribs ,sternum and aerated lungs had been considered obstacles to ultrasound waves (Dietrich C, et al., 2015). However improvements in technology have lead to production of higher-resolution transducers and techniques such as tissue harmonic imaging, which lead to improved spatial resolution and deeper tissue penetration of ultrasound waves (Lameh A et al. ,2019),also the pathological processes as inflammations ,trauma or neoplastic within the chest wall ,pleural, and lungs result in profound changes in tissue composition and improved acoustic transmission and allow for adequate lungs sonographic evaluation(Dietrich C, et al., 2015).

Chest sonography serves as a powerful complementary diagnostic tool with advantage of easy availability ,rapid ,radiation free (Dietrich C, et al., 2015), repeatable and inexpensive methods, determining the high diagnostic accuracy in detecting pediatric chest lesions (Lameh A et al .,2019).

Causes of pediatric chest X ray opacity:

Radio-opacities are more common and significant compared to increased radiolucency , can be caused by many different pathologies and present with different patterns (Gelaw S.,2015), as:

Consolidation:

Caused by replacement of the air in distal airways and the alveoli by fluid or soft tissues. Radiological, this is seen as opacity of any size and mostly homogenous, it has no volume loss, has the tendency to coalescence, has ill-defined margins, non-segmental distribution, irregular shape, air bronchogram (Gelaw S.,2015).

By ultrasound its similar in echogenicity and echotexture to liver and spleen. Bronchograms present within the solid appearing area of echogenicity as multiple bright dot like , and branching linear structures represent air in bronchi and scattered residual air in alveoli(Barillari A et al. ,2011).

Differentiate from atelectasia by presence of dynamic air bronchogram (Barillari A et al .,2011).

Collapse (atelectasis):

This may affect the whole hemi-lung or sub-division of the lungs, such as the lobes , segments or subsegments of the lung. Radiological, it causes opacity and signs of volume loss(Gelaw S.,2015).

It is important to to differentiate focal areas of cosolidation from those of collapse ,since collapse may be associated with a foreign body inhalation or other extrinisic obstruction (Arthur R.,2003) . By chest ultrasound atelectasis similar in echogenicity and echotexture to liver and the air broncograms appear crowded and parallel (Barillari A et al.,2011).

Interstitial opacities:

This is the common presentation of chronic diffuse interstitial lung diseases (Gelaw S.,2015).

Lung ultrasound is an emerging tool in diagnosis of interstitial lung diseases by evaluation number of B lines ,pleural irregularities and nodules or consolidation (Falcetta et al., 2018).

Pleural/chest wall opacities:

Pleural opacities, such as pleural mass lesion, pleural thickening or calcification or mass arising from soft tissue or bony chest wall (Gelaw S., 2015) , in the pleural effusion is challenging to differentiate between the pleural effusion and consolidation by the X ray especially in hemithorax (Prina E., 2014).ultrasound provides detailed information about the nature of pleural fluid and allows one to determine whether a fluid collection is amenable to aspiration (Kim O et al., 2000).

Nodular opacities or mass:

These are rounded increased opacities that can be caused by different pathologies. Radiological , these can be seen on any location, with sizes ranging from pinpoint to mass (it is called mass if >3 cm), solitary or multiple (such as miliary nodules, if multiple small nodules ≈2 mm in diameter), can have different shapes; and margins can be smooth, umbilicated or lobulated. The outline can be sharp, ill-defined or speculated (Gelaw S.,2015).

Ring opacities:

These are annular opacities with central radiolucency usually due to cavitations of pre-existing lesion, but also can be caused by bullae, benign air cyst, loculated pneumothorax or fibrocystic changes (Gelaw S.,2015).

Linear opacities:

These are thin or thick (band shadow, if 5 mm or more) linear shadows. The most common abnormal linear opacity is a scar. Post-primary tuberculosis commonly heals with fibrosis presenting with irregular linear opacities with or without volume loss (Gelaw S.,2015).

ELIGIBILITY:
Inclusion Criteria:

* Age more than twenty eight day up to 18 yrs .

  * Patients admitted in ER &chest wards ,with history of fever cough and dyspnea .
  * Chest X ray opacity on recent admission .
  * Patients who developed acute chest infection on top of chronic respiratory disease .

Exclusion Criteria:

* • Neonate .

  * Chronic disease as cardiac disease

Ages: 29 Days to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: The pediatric patients admitted in ER &chest wards in Assiut University Children Hospital .
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Value of Chest Ultrasound in Detecting causes of Radiological Opacities in Comparison to CT scan Among Children at Assiut University Children Hospital | baseline
  To evaluate the accuracy of chest ultrasound for diagnosis of different lung lesions in comparison to the gold standard among children

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Hassan, professor, Study Director — Assiut University; Yasser Rezk, Lecturer, Study Director — Assiut University; Mohamed Aboelela, Lecturer, Study Director — Assiut University; Sahar Youssif, Lecturer, Study Director — Assiut University